CLINICAL TRIAL: NCT06025604
Title: Psycho Social Factors Associated to Return to Work After Breast Cancer Care : a Prognostic Study
Brief Title: ACTIVPROSEIN : Professional Activity After Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC23.0151; 2023-A01036-39 (Other: ID RCB)
Record Dates: First submitted 2023-07-27; First posted 2023-09-06 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer Female; Return to Work
Keywords: Observational study; Prognostic factors; Questionary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer is, in term of incidence, the first cancer among women in France and worldwide. This incidence is increasing, particularly among young women during their professional activity.

Those observations raise de question of return to work of those patients, and, broadly, of the post cancer life and former activities recovery.

The objective of the study is to identify any factor influencing time from diagnosis to return to work (type of treatment, side effects, residual symptoms, medical staff support, occupational physician monitoring, individual or group supportive therapy, adapted physical activity, alternative therapeutics ..), and the main modalities of return to work (part or full time, professional redeployment).

To identify those factors, barriers or supports, would enable the implementation of concrete actions and programs, promoting return to work, and to a free disease life for those patients.

The main objective is to identify psycho social factors involved in the time from diagnosis to return to any modality of work, until 24 month after localized breast cancer care, in Grenoble University Hospital (Michalon and Voiron included) Secondary objectives are to identify psycho social factors involved in the time from diagnosis to return to work, part time, full time, and redeployment, respectively, until 24 month after localized breast cancer care, in Grenoble University Hospital (Michalon and Voiron included)

DETAILED DESCRIPTION:
Patients being took care in Grenoble University Hospital, including Voiron site, from 2015 to 2019, for a localized breast cancer, will be identified be Cristal Link software.

A questionary, including every studied variables and potential confounding factors, will be sent, by post or by e mail, to the patients. An information notice and a non opposition formulary will be joined to the questionary.

Patients will be contacted by a paramedical member of the Women Cancer Center of the University Hospital, in order to explain them the objective of the study, and the modality of personal data management.

The questionary will be returned either by mail, or directly brought back to the Hospital along a medical appointment.

Data collection will focus on return to work delay, return to work modality (part or full time, redeployment), studied variables and potential confounding factors (demographic : marital status, number of dependent children, incomes / related to occupational activity : night work, job responsibility, occupational physician follow up / treatment consequences : OMS status, anxiety, depression, lymphoedema, articular pain, neuropathic pain / Support measures : physical activities, psychological support, alternative therapeutics, familial support, medical staff support).

Medical data (tumour features : histology, extent, treatment : surgery, chemiotherapy, targeted therapy, hormonotherapy, radiotherapy) will be collected using informatic files.

Subjective variables will be evaluated using standardized questionary (Anxiety : Stait Trait Anxiety Inventory / Depression : Hamilton Depression Scale / Cognition : FACT cog questionary / Support : Multidimensional Scale of Support).

Data process will be done in the Clinical Investigation Center of Grenoble University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 60 years old
* Histologically proven localized breast cancer, of any subtype
* Cared in Grenoble University Hospital between 2015 and 2019
* Working at the time of diagnosis

Exclusion Criteria:

* Retired at the end of adjuvant therapy
* Deprived of liberty, under juridical protection, not able to give consent
* Psychiatric conditions or addictive behavior interfering with questionary filling

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Women between 18 and 60 years old, care in Grenoble University Hospital between 2015 and 2019 for a localized breast cancer, working at the time of diagnosis.
Sampling Method: Probability Sample
Enrollment: 578 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-09-13 (Estimated); Study Completion 2025-09-13 (Estimated)

PRIMARY OUTCOMES:
To identify the impact of psycho social factors on delay of return to any modality of work, until 24 months after localized breast cancer care, in Grenoble University Hospital (Michalon and Voiron included) | 30 minutes
  Assessment of delay of a any occupational activity recovery, from the diagnosis and until 24 months after treatment, and of any influenced factors by self administrated questionnaire, included standardized questionnaire for subjective variables

SECONDARY OUTCOMES:
To identify the impact of psycho social factors on delay of return to full time work, until 24 months after localized breast cancer care, in Grenoble University Hospital (Michalon and Voiron included) | 30 minutes
  Assessment of delay of full time work recovery, from the diagnosis and until 24 months after treatment, and of any influenced factors by self administrated questionnaire, included standardized questionnaire for subjective variables
To identify the impact of psycho social factors on delay of return to part time work, until 24 months after localized breast cancer care, in Grenoble University Hospital (Michalon and Voiron included) | 30 minutes
  Assessment of delay of part time work recovery, from the diagnosis and until 24 months after treatment, and of any influenced factors by self administrated questionnaire, included standardized questionnaire for subjective variables
To identify the impact of psycho social factors on delay of return to occupational reclassification, until 24 months after localized breast cancer care, in Grenoble University Hospital (Michalon and Voiron included) | 30 minutes
  Assessment of delay of occupational reclassification, from the diagnosis and until 24 months after treatment, and of any influenced factors by self administrated questionnaire, included standardized questionnaire for subjective variables

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, Grenoble, France